CLINICAL TRIAL: NCT05836324
Title: A Phase 1, Open-Label, Multicenter Study of INCA33890 in Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety of INCA33890 in Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCA 33890-101; 2022-502456-31-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-04-14; First posted 2023-05-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors; Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Solid Tumors; INCA33890
MeSH Terms: interventions — Bevacizumab; IFL protocol; Folfox protocol; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1a - Dose Escalation Monotherapy (Experimental): INCA33890 will be administered at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890
- Part 1b-Dose Expansion Monotherapy (Experimental): INCA33890 will be administered at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890
- Part 2a - Dose Escalation Combination Therapy - Group 1 (Experimental): INCA33890 will be administered in combination with bevacizumab at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: bevacizumab
- Part 2a - Dose Escalation Combination Therapy - Group 2 (Experimental): INCA33890 will be administered in combination with bevacizumab and FOLFIRI at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: bevacizumab; Drug: FOLFIRI
- Part 2a - Dose Escalation Combination Therapy - Group 3 (Experimental): INCA33890 will be administered in combination with bevacizumab and FOLFOX at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: bevacizumab; Drug: FOLFOX
- Part 2a - Dose Escalation Combination Therapy - Group 4 (Experimental): INCA33890 will be administered in combination with cetuximab at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: Cetuximab
- Part 2b - Dose Expansion Combination Therapy - Group 1 (Experimental): INCA33890 will be administered in combination with bevacizumab at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: bevacizumab
- Part 2b - Dose Expansion Combination Therapy - Group 2 (Experimental): INCA33890 will be administered in combination with bevacizumab and FOLFIRI at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: bevacizumab; Drug: FOLFIRI
- Part 2b - Dose Expansion Combination Therapy - Group 3 (Experimental): INCA33890 will be administered in combination with bevacizumab and FOLFOX at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: bevacizumab; Drug: FOLFOX
- Part 2b - Dose Expansion Combination Therapy - Group 4 (Experimental): INCA33890 will be administered in combination with cetuximab at the protocol-defined dose based on cohort assignment.
  Interventions: Drug: INCA33890; Drug: Cetuximab

INTERVENTIONS:
Drug: INCA33890 — INCA33890 will be administered at protocol defined dose.
Drug: bevacizumab — Bevacizumab will be administered at protocol defined dose.
  Arms: Part 2a - Dose Escalation Combination Therapy - Group 1; Part 2a - Dose Escalation Combination Therapy - Group 2; Part 2a - Dose Escalation Combination Therapy - Group 3; Part 2b - Dose Expansion Combination Therapy - Group 1; Part 2b - Dose Expansion Combination Therapy - Group 2; Part 2b - Dose Expansion Combination Therapy - Group 3
Drug: FOLFIRI — FOLFIRI will be administered at protocol defined dose.
  Arms: Part 2a - Dose Escalation Combination Therapy - Group 2; Part 2b - Dose Expansion Combination Therapy - Group 2
Drug: FOLFOX — FOLFOX will be administered at protocol defined dose.
  Arms: Part 2a - Dose Escalation Combination Therapy - Group 3; Part 2b - Dose Expansion Combination Therapy - Group 3
Drug: Cetuximab — Cetuximab will be administered at protocol defined dose.
  Arms: Part 2a - Dose Escalation Combination Therapy - Group 4; Part 2b - Dose Expansion Combination Therapy - Group 4

SUMMARY:
To evaluate the safety, tolerability, and DLTs and determine the MTD and/or RDE(s) of INCA33890 in participants with select advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Histologically or cytologically confirmed advanced or metastatic malignancies as defined in the protocol.
* Part 1: Participants must have experienced disease progression after treatment with, be intolerant to, or be ineligible for, or refused available therapies, including anti-PD-(L)1 or anti-CTLA4 therapy if applicable, that are known to confer clinical benefit. Part 2: depending on cohort, participants may have received or not prior treatment for the malignancy under study.
* ECOG performance status score of 0 or 1.
* Willingness to undergo pre- and on-treatment tumor biopsy (core or excisional). Biopsies are mandatory depending on the cohorts.
* Presence of measurable disease according to RECIST v1.1.

Exclusion Criteria:

* Any known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years.
* Not recovered to ≤ Grade 1 or baseline from residual toxicities of prior therapy.
* Has active autoimmune disease requiring systemic immunosuppression with corticosteroids.
* Brain or CNS metastases untreated or that have progressed.
* History of organ transplant, including allogeneic stem cell transplantation.
* History of clinically significant or uncontrolled cardiac disease.
* Active HBV, active HCV, or HIV positive.
* Is on chronic systemic steroids (> 10 mg/day of prednisone or equivalent).
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment
* Participants that have been initiated on or had modifications in anticoagulation therapies within the last 3 months prior to first dose of treatment.
* Significant concurrent, uncontrolled medical condition, eg:

  * Cardiovascular: Participants with known vasculitis, aneurisms, and other vascular malformations of clinical significance or history of myocarditis.
  * Gastrointestinal: Any bowel obstruction within 60 days prior to C1D1.
* Participants with adequate laboratory values within the protocol defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-01-13 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | Up to 28 days
Treatment Emerging Adverse Events (TEAEs) | Up to 2 years
TEAEs leading to dose modification or discontinuation | Up to 2 years

SECONDARY OUTCOMES:
Objective response Rate | 2 years
Disease Control Rate | 2 years
Duration of Response | 2 years
Pharmacokinetics Parameter : Cmax of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up
Pharmacokinetics Parameter : Tmax of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up
Pharmacokinetics Parameter : Cmin of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up
Pharmacokinetics Parameter : AUC(0-t) of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up
Pharmacokinetics Parameter : AUC 0-∞ of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up
Pharmacokinetics Parameter : CL of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up
Pharmacokinetics Parameter : Vz of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up
Pharmacokinetics Parameter : t1/2 of INCA33890 | Pre dose - Day 1 of Cycle 1(C1D1)- 28 (each cycle is 28 days), Day 15 of Cycle 1-3; 10min and 4hrs Post dose(PD) - C1D1,C1D4, 24hrs PD C1D2, any time PD Day 4, 8, 22, of Cycle 1, and any time during 30 day Follow Up

CONTACTS AND LOCATIONS:
Locations (36):
- United States (11):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer and Hematology Centers of Western Michigan-Start Midwest, Grand Rapids, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Nyu Langone Health - Long Island Hospital, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lifespan Cancer Research Institute, Providence, Rhode Island
  - University of Texas Md Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Denmark (4):
  - Rigshospitalet Uni of Hospital of Copenhagen, Copenhagen
  - Herlev Og Gentofte Hospital, Herlev
  - Odense University Hospital, Odense C
  - Vejle Hospital, Vejle
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Centro Ricerche Cliniche Di Verona, Verona
- Japan (3):
  - Kansai Medical University Hospital, Hirakata
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Jfcr, Tokyo
- Spain (5):
  - Start Barcelona, Barcelona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
- Switzerland (3):
  - Istituto Oncologico Della Svizzera Italiana, Bellinzona
  - Centre Hospitalier Universitaire Vaudois (Chuv), Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (5):
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - Guys and St Thomas Nhs Foundation Trust, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - Freeman Hospital Newcastle Upon Tyne Foundation Nhs Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study to evaluate the safety of INCA33890 in Participants With Advanced or Metastatic Solid Tumors — https://incyteclinicaltrials.com/studies/inca-33890-101